CLINICAL TRIAL: NCT00973336
Title: Primary Hyperparathyroidism: Does a Systematic Treatment Improve the Calcium and Bone Metabolism After Successful Surgery in Patients Without Osteoporosis?
Brief Title: Primary Hyperparathyroidism: Does a Systematic Treatment Improve the Calcium and Bone Metabolism After Surgery?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Philipp Riss, Assistent Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHPT02_2008
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Primary Hyperparathyroidism; Bone Metabolism
Keywords: postoperative follow-up
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Calcium; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium and vitamin D (Experimental): Intervention
  Interventions: Drug: Calcium and vitamin D
- No treatment (control) (No Intervention)

INTERVENTIONS:
Drug: Calcium and vitamin D — 1000mg calcium per day 800 IE vitamin D per day
  Arms: Calcium and vitamin D

SUMMARY:
Primary Hyperparathyroidism (pHPT) increases bone turnover and resorption and thus calcium efflux out of bone. After successful surgical treatment of pHPT, bone takes up calcium again which may result in secondary hyperparathyroidism or even "hungry bone syndrome". Until today there are no studies about this problem helping to develop recommendations or guidelines how to prevent these symptoms.

Study hypothesis: Calcium and vitamin D intake after surgery for PHPT protects the bone by keeping PTH in the normal range (less secondary, reactive hyperparathyroidism), prevents hungry bone- syndrome and improve bone-turnover markers (osteoporosis protection).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Male patients
* Biochemically proven PHPT, PTX planned
* No evidence for osteoporosis

Exclusion Criteria:

* Postoperative hypocalcemia needing substitution with calcium and vitamin D/ 1-25-OH-Vitamin D
* Cancer (lung, breast, prostatic, parathyroid cancer and thyroid carcinoma >1cm)
* Persisting or recurrent PHPT (postoperative hypercalcemia)
* Four-gland hyperplasia
* Multiple endocrine neoplasia (MEN) or hereditary PHPT
* Familial hypercalciuric hypercalcaemia (Ca/creatinine ratio < 0.01)
* Phenylketonuria
* Renal impairment (creatinine clearance <30ml/h)
* Severe hepatic disorder
* Severe systemic disorder
* Thyroid dysfunction
* Immobilisation
* Intake of drugs with potential effects on BMD like glucocorticoids, lithium, estrogen-replacement therapy, selective Estrogen-receptor modulators (sERMs), bisphosphonates in the last three months
* Intake of drugs containing digoxin or digitoxin
* Known allergy against any component of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Parathyroid hormone | 1 year

SECONDARY OUTCOMES:
BMD of lumbar spine, femoral neck and radius | 1 year
Adverse effects calcium or vitamin D | 1 year
Other biochemical markers of bone metabolism | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Niederle, Prof., MD, Principal Investigator — Medical University of Vienna, Department of Surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria